CLINICAL TRIAL: NCT04967898
Title: Comparison of Bowen Technique and Sustain Stretching on Hamstring Flexibility in Asymptomatic Females
Brief Title: Effect of Manual Technique on Hamstring Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/Lhr/20/0112 Mahnoor
Record Dates: First submitted 2021-07-19; First posted 2021-07-20 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Muscle Tightness
Keywords: sit and reach test, Bowen technique

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bowen technique (Experimental): group 1 will be treated with the Bowen technique and heating pad. this technique will be given to asymptomatic females. 22 subjects will be taken this treatment. treatment will be given thrice a week for 3 weeks. the subjects will come after 1 month for follow-up.
  Interventions: Other: bowen technique
- sustained stretching (Active Comparator): group 1 will be treated with the sustained stretching technique and heating pad. this technique will be given to asymptomatic females. 22 subjects will be taken this treatment. treatment will be given thrice a week for 3 weeks. the subjects will come after 1 month for follow-up
  Interventions: Other: sustained stretching

INTERVENTIONS:
Other: bowen technique — Bowen technique is a soft tissue mobilization technique. This medical care involves short mild rolling moves over the muscles, nerves, ligaments, and tendons of flesh utilizing the hands, fingers and thumb. Sequence of receiving bilateral rolling moves over segments of the erector spinae from the lumber toward cervical spine, latissimus dorsi, the gluteal, the hamstring muscles proximally and distally, tensor facia Lata and a medial hip striated muscle move.
  Arms: bowen technique
Other: sustained stretching — static stretching is one of the most common and safest technique used for hamstring tightness. A static stretch is performed by inserting muscles at their greatest attainable length and holding that position for an amount of your time.
  Arms: sustained stretching

SUMMARY:
This study will be a randomized clinical trial. the study will be conducted in Mubarak Hospital Sargodha. a sample size of 44 subjects will be taken. subjects will be divided into two groups using the lottery method. group 1 will be treated with Bowen technique along with heating pad and group 2 will be treated with sustained stretching technique along with heating pads thrice a week for 3 weeks. subjects will come after 1 month for follow up. the follow-up will show which technique is more effective in improving hamstring flexibility and range in healthy females. the outcome measures active knee extension test and sit and reach test will be used to check hamstring flexibility and range at baseline, post-treatment, and follow-up. data were analyzed using spss 26.

DETAILED DESCRIPTION:
hamstring muscles are responsible for hip and knee movement during walking, running, squatting, bending knees, and pelvis tilting. hamstring muscles function is to perform flexion at knee and hip extension. hamstring tightness is more common in females than males. once the hamstring were tightened ,incidence of low back pain rose to 15%.

hamstring shortening occurred due to maintain same posture for prolong period of time, fatigue, sedentary life style, and poor body mechanics. hamstring tightness can disturb the biomechanics of low back and pelvis in each adolescents and adult. most of the individuals with hamstring tightness were asymptomatic. Throughout daily activities, nerves that innervate the hamstring muscle is exposed to constant pressure throughout sitting, standing can cause hamstring tightness.. Nerve adhesions inside the hamstring may alter neurodynamic inflicting abnormal machan-o-sensitivity of the nerve that will influence hamstring flexibility. This machan-o-sensitivity of the neural tissue could limit hamstring length in traditional healthy people. Shortened hamstrings amendment the curvature of the spine inflicting larger compression masses within the mesial curvatures and increase in intradiscal pressure and also the incidence of larger shear forces, thereby predisposing people to spinal issues various techniques were used to treat hamstring tightness. this study we compare the effects of Bowen technique and sustained stretching on hamstring flexibility in asymptomatic females.

group 1 will be treated with Bowen technique .this is a soft tissue mobilization technique This medical care involves short mild rolling moves over the muscles, nerve, ligaments and tendons of flesh utilizing the hands, fingers and thumb. Sequence of receiving bilateral rolling moves over segments of the erector spinae from the lumber toward cervical spine, latissimus dorsi, the gluteal, the hamstring muscles proximally and distally, tensor facia Lata and a medial hip striated muscle move. Treatment will be given thrice a week for 3 weeks. and treatment session will be 20minutes for each leg.

group 2 will be treated with sustained stretching technique. Sustained stretching is most common and safest technique used for hamstring tightness. This sort of stretch is applied slowly and bit by bit at a comparatively constant force to avoid eliciting a inborn reflex. The resultant increase in muscle length is said to elastic behavior. Static stretch of thirty seconds at a frequency of 3 continual stretches per single session is ample to extend muscle length. treatment will be given thrice a week for 3 weeks. Treatment session will be 30 seconds for each leg. both groups will come after 1 month for follow up. Outcome measure active knee test and sit and reach test will be used to check hamstring flexibility and range in asymptomatic females at baseline, post-treatment and follow up. the goal of this study is to improve hamstring flexibility in asymptomatic females.

active knee extension test and sit and reach test will be used to check hamstring flexibility and range in subjects. these both tests have very high reliability and validity. There is a lack of evidence demonstrating the effects of Bowen technique and sustained stretching on hamstring flexibility. the purpose of this study is to compare the effects of both techniques to assess which technique has more clinical impact than other.

ELIGIBILITY:
Inclusion Criteria:

* age 25-40 years
* asymptomatic subjects
* both hamstring tightness
* only females

Exclusion Criteria:

* females with past history of hamstring tightness
* previous surgery
* pathology
* female with back pain and spinal deformity

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female 25-40 years
Enrollment: 44 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
active knee extension test | 3 weeks
  Active Knee Extension test (AKE) or Popliteal angle test or 90/90 test: This test was found as gold standard test for estimating hamstring flexibility. This test is used to assess the hamstring muscle length and range of active knee extension with hip in flexed position.
sit and reach test | 3 weeks
  Sit and reach test is a common measure of flexibility. This test help to measure the extensibility of hamstring and lower back.
  super > +27 > +10.5 > +30 > +11.5 excellent +17 to +27 +6.5 to +10.5 +21 to +30 +8.0 to +11.5 good +6 to +16 +2.5 to +6.0 +11 to +20 +4.5 to +7.5 average 0 to +5 0 to +2.0 +1 to +10 +0.5 to +4.0 fair -8 to -1 -3.0 to -0.5 -7 to 0 -2.5 to 0 poor -20 to -9 -7.5 to -3.5 -15 to -8 -6.0 to -3.0 very poor < -20 < -7.5 < -15 < -6.0

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Mubarak Hospital, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marr M, Baker J, Lambon N, Perry J. The effects of the Bowen technique on hamstring flexibility over time: a randomised controlled trial. J Bodyw Mov Ther. 2011 Jul;15(3):281-90. doi: 10.1016/j.jbmt.2010.07.008. Epub 2010 Sep 15. PMID 21665103
- [Background] Meroni R, Cerri CG, Lanzarini C, Barindelli G, Morte GD, Gessaga V, Cesana GC, De Vito G. Comparison of active stretching technique and static stretching technique on hamstring flexibility. Clin J Sport Med. 2010 Jan;20(1):8-14. doi: 10.1097/JSM.0b013e3181c96722. PMID 20051728
- [Background] Starring DT, Gossman MR, Nicholson GG Jr, Lemons J. Comparison of cyclic and sustained passive stretching using a mechanical device to increase resting length of hamstring muscles. Phys Ther. 1988 Mar;68(3):314-20. doi: 10.1093/ptj/68.3.314. PMID 3347651
- [Background] Medeiros DM, Cini A, Sbruzzi G, Lima CS. Influence of static stretching on hamstring flexibility in healthy young adults: Systematic review and meta-analysis. Physiother Theory Pract. 2016 Aug;32(6):438-445. doi: 10.1080/09593985.2016.1204401. Epub 2016 Jul 26. PMID 27458757
- [Background] Shadmehr A, Hadian MR, Naiemi SS, Jalaie S. Hamstring flexibility in young women following passive stretch and muscle energy technique. J Back Musculoskelet Rehabil. 2009;22(3):143-8. doi: 10.3233/BMR-2009-0227. PMID 20023343